CLINICAL TRIAL: NCT04982458
Title: Clinical Study of 68 GA-FAPI PET Imaging Noninvasive Visible Fibrosis Formation in Heart Failure
Brief Title: Visualized Monitoring of Fibrosis Formation in Heart Failure With 68GA-FAPI PET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan-0617-01
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Positron Emission Tomography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI — 68Ga-FAPI injection is a radiopharmaceutical used for positron emission tomography (PET) diagnosis. This product is used for PET, qualitative and localized diagnosis and evaluation of abnormal expression of fibroblast-activated protein in focus-associated fibroblasts.

SUMMARY:
This is a diagnostic study. Patients were included from patients with clinically suspected or confirmed heart failure, and 68Ga-FAPI and 13N-NH3 gated myocardial imaging were performed to evaluate the effectiveness of 68Ga-FAPI PET imaging in visualizing the degree of myocardial fibrosis in patients with heart failure. The subjects completed 68Ga-FAPI and 13N-NH3 gated myocardial imaging in a one-stop process, and collected general information, clinical data, echocardiography, blood routine, liver and kidney function indicators, 68Ga-FAPI and 13N-NH3 PET imaging results and other imaging data of the patients and volunteers.

DETAILED DESCRIPTION:
Fibroblast activated protein (FAP) is a type II membrane-bound glycoprotein that is highly specifically expressed in activated fibroblast reactions. The 68Ga labeled fibroblast activated protein inhibitor (68 ga-fapi) has shown advantages of high uptake and high image contrast in imaging the activated fibroblast response, including its successful use in visualizing the degree of liver fibrosis. The molecular imaging probe targeting FAP combined with the mature myocardial perfusion imaging agent 13N-NH3 can help us to achieve the following objectives: On the one hand, to investigate the myocardial fibrosis in patients with heart failure and to visualize the formation of fiBER-activated protein in the process of heart failure; At the same time, the performance of 68GA-FAPI in differential diagnosis of heart failure and grading of heart failure degree was discussed, so as to make up for the insufficiency of clinical routine imaging technology in the diagnosis of myocardial fibrosis in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or above), gender is not limited;
* Patients with clinically suspected or confirmed heart failure (supporting evidence includes visual examination, cardiac MRI, cardiac ultrasound, and serological indicators, etc.), and patients who agree to undergo 68Ga-FAPI and 13N-NH3 imaging;
* The patient or his legal representative can sign the informed consent.

Exclusion Criteria:

* Acute systemic diseases and electrolyte disorders；
* Pregnant or lactating women；
* Patients refuse to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected or confirmed heart failure (supporting evidence including visual examination, cardiac MRI, cardiac ultrasound, and serological indicators, etc.), and who have consenting to 68GA-FAPI and 13N-NH3 imaging;
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga-FAPI PET for diagnosis and staging in heart failure. | 2 years
  For 50 subjects with suspected or diagnosed or treated heart failure who have completed 13N-NH3 imaging, diagnosis and staging results of 68Ga-FAPI PET will be compared to pathology, clinical and follow-up result.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Xiaoli Lan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song W, Zhang X, He S, Gai Y, Qin C, Hu F, Wang Y, Wang Z, Bai P, Wang J, Lan X. 68Ga-FAPI PET visualize heart failure: from mechanism to clinic. Eur J Nucl Med Mol Imaging. 2023 Jan;50(2):475-485. doi: 10.1007/s00259-022-05994-4. Epub 2022 Oct 21. PMID 36269382